CLINICAL TRIAL: NCT02056821
Title: Hemodynamic Effects on Cerebral Autoregulation in Acute Stroke
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, Joseph Miller, MD, Senior Staff, Henry Ford Health System
Other Study IDs: A20030
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Ischemic Stroke
Keywords: stroke; transcranial doppler; cerebral blood flow; cardiac output; non-invasive hemodynamic monitoring
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates if there are hemodynamic alterations in acute stroke that predispose patients to impaired perfusion and regulation of cerebral blood flow. To test this, we will target recruitment of acute ischemic stroke patients who present to the ED within 12 hours of symptoms onset. Enrolled subjects will receive continuous noninvasive hemodynamic monitoring contemporaneous with measurements of cerebral blood flow velocities and cerebral oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Suspected ischemic stroke within 12 hours of symptom onset
* NIHSS ≥ 4
* Age 18 to 90 years

Exclusion Criteria:

* Baseline modified Rankin Scale > 3
* Pregnancy
* Intracranial hemorrhage on head CT
* Mechanical ventilation prior to enrollment
* Inadequate temporal windows for TCD analysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute (< 12 hours) ischemic stroke patients presenting to the Emergency Department
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow velocities | initial 24 hours
  Cerebral flow velocities determined by bilateral MCA measurements by TCD

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Derived] Miller J, Moloney JA, Elagamy N, Tuttle J, Tirgari S, Calo S, Thompson R, Nahab B, Lewandowski C, Levy P. Cerebral blood flow change with fluid resuscitation in acute ischemic stroke. Brain Circ. 2024 Dec 28;10(4):303-307. doi: 10.4103/bc.bc_30_24. eCollection 2024 Oct-Dec. PMID 40012591